CLINICAL TRIAL: NCT00105768
Title: Effectiveness of Advisor - Teller Money Manager (ATM)
Brief Title: Effectiveness of Advisor-Teller Money Manager
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHI 20-001
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-03

CONDITIONS: Substance Abuse; Dual Diagnosis
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Advisor-Teller Money Management-Substance Abuse Counselling

INTERVENTIONS:
Behavioral: Advisor-Teller Money Management-Substance Abuse Counselling

SUMMARY:
VA investigators have described greater substance use at the beginning of the month when disability and other monthly checks are received. The proposed research addresses an important VA priority�seeing that veterans� funds are spent to improve veterans� quality of life and are not misspent on substances of abuse.

DETAILED DESCRIPTION:
Background:

VA investigators have described greater substance use at the beginning of the month when disability and other monthly checks are received. The proposed research addresses an important VA priority�seeing that veterans� funds are spent to improve veterans� quality of life and are not misspent on substances of abuse.

Objectives:

The objective was to determine the effectiveness of a money management-based therapy called ATM for veterans who abuse cocaine or alcohol compared to a financial advice control condition.

Methods:

Veterans were randomly assigned to 36-weeks of ATM or to the control condition, financial advice. ATM (Adviser-Teller Money Manager) involves meeting with a money manager at least weekly. The money manager performs three functions�limiting patients� access to funds by storing checkbooks and ATM cards, training patients to budget their funds, and linking spending to treatment goals. The control condition involved listing income and expenses in a workbook. Veterans were enrolled from each of two sites if they had spent at least $100 in the preceding 90 days on alcohol or cocaine, and had at least $300 per month income. Measures of treatment fidelity and participation included number of visits attended, whether funds were stored, monthly income and expenses and Likert-scaled ratings from 1-4 of money management-related outcomes. Outcome measures collected included urine toxicology tests and breathalyzers, self-reported substance use as assessed by the ASI follow-up, and secondary measures including quality of life and psychiatric symptomatology.

Status:

Data analysis is ongoing. Attempts are being made to (a) disseminate ATM and assess its effect among homeless women veterans (b) determine the reliability and validity of money management-based assessments used to determine which veterans are capable of managing their funds (c) optimize funds management by disabled veterans.

ELIGIBILITY:
Inclusion Criteria:

Age _>18. Meets DSM-II criteria for cocaine abuse or alcohol abuse. Self-reported use of at least $100 worth of alcohol or cocaine during 30 days within last 90 days. Income of at least $300 per month.

Exclusion Criteria:

Currently receives money management, physiological dependence on alcohol or opiates, has a conservator or other payee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2002-07; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Weeks of abstinence

SECONDARY OUTCOMES:
Participation in the Intervention, Service Use, Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Marc I. Rosen, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

REFERENCES:
- [Result] Rosen MI, Bailey M, Rosenheck RR. Alcohol & drug abuse: principles of money management as a therapy for addiction. Psychiatr Serv. 2003 Feb;54(2):171-3. doi: 10.1176/appi.ps.54.2.171. No abstract available. PMID 12556596
- [Result] Rosen MI, Rosenheck R, Shaner A, Eckman T, Gamache G, Krebs C. Do patients who mismanage their funds use more health services? Adm Policy Ment Health. 2003 Nov;31(2):131-40. doi: 10.1023/b:apih.0000003018.16515.32. PMID 14756196
- [Result] Black RA, Rounsaville BJ, Rosenheck RA, Conrad KJ, Ball SA, Rosen MI. Measuring money mismanagement among dually diagnosed clients. J Nerv Ment Dis. 2008 Jul;196(7):576-9. doi: 10.1097/NMD.0b013e31817d0535. PMID 18626300